CLINICAL TRIAL: NCT00633958
Title: A Pilot, Non-Therapeutic NeuroImaging Study of 18F-FLT in Pediatric Patients With Newly Diagnosed Central Nervous System Tumors
Brief Title: A Pilot Study of 18F-FLT in Pediatric Patients With Central Nervous System (CNS) Tumors
Acronym: FLT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Large phase II opened to accue same patients
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 05-303
Record Dates: First submitted 2008-03-05; First posted 2008-03-12 (Estimated); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Tumors of the Central Nervous System
Keywords: 18F-FLT; FLT; PET; CNS tumors; Newly; diagnosed
MeSH Terms: conditions — Central Nervous System Neoplasms; Disease | interventions — alovudine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- 18F-FLT (Experimental): All subjects will receive 18F-FLT prior to PET imaging.
  Interventions: Drug: 18F-FLT; Radiation: PET Imaging

INTERVENTIONS:
Drug: 18F-FLT — Patients will receive a dose of 18F-FLT through a fresh intravenous catheter as per standard PET procedures. Dosing will be based on age.
  Other Names: 18F]-Fluorothymidine
Radiation: PET Imaging

SUMMARY:
In spite of numerous advances in neuroimaging techniques, the diagnosis of pediatric brain tumors relies on the pathologic evaluation of material obtained at the time of the initial operation. While 18F-FDG-positron emission tomography (PET) helps identify higher-grade lesions due to their increased glucose metabolism, the high tracer uptake of the normal adjacent brains makes this modality of limited value. Fluorine-18 fluorothymidine (FLT) is a new imaging agent that has two significant advantages in the imaging of CNS tumors. First, this agent detects cellular proliferation directly, and second, the normal brain does not take up the agent, making a positive area(s) easy to identify. Before embarking on a large pediatric disease stratified assessment of FLT imaging in pediatric neurooncology patients, the investigators are proposing a limited patient pilot study to evaluate the biodistribution, dosimetry and specificity of this compound when compared to immunohistochemical assessment of mitotic activity in newly diagnosed patients undergoing surgical resection.

DETAILED DESCRIPTION:
Patients will undergo standard pre-diagnostic imaging of the sites of disease using standard MRI techniques. If disease is suspected in both the brain and spine, then both imaging modalities should be obtained. This imaging should be obtained no more than 21 days before surgical resection. As close as possible to the completion of the MRI scans, patients will undergo 18F-FLT imaging using a single administration of tracer, and PET image acquisition at four different time points (baseline, 1 hr post injection, 2 hrs post injection and 4-6 hours post injection). A whole body PET scan (top of the head to mid thigh) will be performed immediately after injection (PET acquisition #1). These data will be acquired with a 2 minute emission and a 2 minute transmission scan at each bed position. Following this acquisition, the subject will empty his or her bladder. At 45 minutes post-injection, a brain and/or spine (body) PET scan will be acquired with a 10 min emission scan and a 5 min transmission scan (PET acquisition #2). This scan will include all areas of suspected tumor (brain, spine, or brain and spine). Following PET acquisition #2, a whole body PET scan will be acquired according to the same protocol as above (PET acquisition #3). If possible, a final whole body scan will be acquired 4-6 h post-injection (PET acquisition #4). All PET acquisitions will be acquired in 3D mode and reconstructed with the FORE re-binned OSEM algorithm with measured attenuation correction. Blood samples will be obtained at the completion of each whole body scan. Patients will receive the dose of 18F-FLT through a fresh intravenous catheter as per standard PET procedures. Patients will then undergo maximal surgical resection. Pieces from different areas of the tumor will be marked for correlation to imaging studies when possible. Tumor samples will undergo standard immunohistochemical analysis for cellular activation including mitotic index and MIB-1 proliferation staining.

Serial blood draws will also be obtained at four different time points (baseline, 1 hr post injection, 2 hrs post injection, and 4-6 hours post injection) to evaluate clearance of 18F-FLT from the blood.

For the biodistribution, the 3D regions of interest (ROIs) will be drawn about each major organ that is identified on the whole body scans. This will be performed on each of the whole body scans and a time activity curve will be generated. The residence time for each organ will be determined. The blood data will be pipetted and counted for estimates of activity in the blood and bone marrow. For the brain and/or spine images, the PET data will be registered to the subjects' MRI. The PET scan will be graded on a subjective 4-point scale. 3D ROIs will be drawn around the tumor. In addition, an analogous ROI will be drawn in normal brain background and about the whole brain for comparison. For the tumor, tumor-to-background, tumor-to-whole brain ratios will be determined. In addition, standard uptake values (SUVs) will be determined for the tumor and background.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with newly diagnosed central nervous system tumors undergoing planned surgical resection within 21 days.
* Patients should be < 21 years of age at the time of diagnosis.
* Patients should be capable of achieving imaging without the need for sedation or anesthesia.
* Karnofsky Performance Status ≥ 50. For infants, the Lansky play scale ≥ 50% can be substituted.
* Patients must not be pregnant or nursing.
* Signed Informed Consent.
* Patients receiving steroids and/or anti-seizure medications are eligible for this study.

Exclusion Criteria:

* Prior radiation therapy and/or chemotherapy are not permitted.
* Active infection
* Pregnancy or breast feeding
* Serious concurrent medical illness

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2008-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To determine the distribution, localization and kinetics of localization of 18F-FLT in pediatric patients with central nervous system tumors | Assessed shortly after subjects undergo neuroimaging

SECONDARY OUTCOMES:
To correlate the activity of administering 18F-FLT in newly diagnosed pediatric brain tumor patients to standard immunohistochemical markers of cellular activation and MRI imaging | Assessed shortly after subjects undergo neuroimaging

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kieran, MD, Principal Investigator — Dana-Farber Cancer Institute/Children's Hospital Boston
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States